CLINICAL TRIAL: NCT01243840
Title: Central Blood Pressure Follow-up Study in Japanese
Brief Title: Japan Central Aortic Pressure Prospective Study
Acronym: J-CARP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yoshio Matsui (Other)
Responsible Party: Sponsor-Investigator, Yoshio Matsui, Sponsor-Investigator, Jichi Medical University
Organization: Jichi Medical University (Other)
Other Study IDs: J-CARP
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Central aortic pressure; Aortic pulse wave velocity; Aortic PWV using a single pressure recording; Vascular aging; Left ventricular hypertrophy; Left ventricular diastolic function
MeSH Terms: conditions — Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose of the study

1. The predictive value of central aortic pressure and aortic pulse wave velocity (PWV) in a Japanese population is not known. The purpose of this study is to quantify the predictive value of these indices in the determination of cardiovascular risk.
2. Recently, a non-invasive method to separate the aortic pressure waveform into the separate ejection pressure wave and reflected pressure wave has become available. With this decomposition method, it is possible to estimate aortic PWV (named AVI). The second objective of this study is to determine if AVI can be a substitute for carotid-femoral PWV (cf-PWV), the current gold standard for aortic PWV measurement.
3. To study vascular aging of the Japanese population by evaluating central blood pressure and aortic PWV by age, and compare these values to similar studies done in Caucasian and Chinese patient populations.
4. To study the relationship between the magnitude of the aortic reflected pressure wave and the degree of left ventricular (LV) hypertrophy and LV diastolic function.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who visit hospital for their health checks
* Healthy volunteers who agree to participate in this study

Exclusion Criteria:

* History of coronary artery disease, cerebrovascular disease, congestive heart failure, aortic dissection
* Subjects taking vasoactive drugs (antihypertensive and/or nitrates)
* Atrial fibrillation or atrial flutter
* Renal dysfunction (serum creatinine ≥3 mg/dl)
* Type I diabetes mellitus
* Hepatic dysfunction (AST and/or ALT ≥100 IU/l)
* A history of malignant tumor within 5 years of enrollment or suspected
* Pregnancy, possible pregnancy
* Chronic inflammation disease
* Not suited to the clinical trial as judged by a collaborating physician
* Inability to give informed consent

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ages eligible for Study: 20 Years to 90 Years Genders eligible for Study: Both Accepts healthy volunteers: Yes
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2010-06; Primary Completion 2014-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
•Composite of following events: sudden death, cardiovascular death, stroke, coronary events, heart failure | 5 years

SECONDARY OUTCOMES:
New onset of hypertension, diabetes mellitus, or atrial fibrillation | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kazuomi Kario, MD, Study Director — Jichi Medical University School of Medicine
Locations (1):
- Iwakuni City Medical Center, Iwakuni, Yamaguchi, Japan